CLINICAL TRIAL: NCT06577896
Title: Safety and Efficacy of 1-month Dual Antiplatelet Therapy in High Bleeding and Ischemic Risk Elderly Patients With Coronary Artery Disease After Implantation of Zotarolimus-eluting Coronary Stent System (Onyx Family, Medtronic, Minneapolis, MN); A Multicenter, Prospective, Observational Study
Brief Title: The Study to Evaluate the Safety and Efficacy of the Onyx Family
Status: Recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Min Ku Chon, Associate Professor, Pusan National University Yangsan Hospital
Other Study IDs: BRONYX STUDY
Record Dates: First submitted 2024-08-27; First posted 2024-08-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Aged 75 or more: Elderly patients aged 75 years or older
  Interventions: Device: Onyx family
- Eligible for interventional procedures: "Patients requiring PCI (Percutaneous Coronary Intervention) procedure
  Interventions: Device: Onyx family
- Evidence of myocardial ischemia or coronary artery stenosis ≥ 50%: Patients with evidence of myocardial ischemia or coronary artery stenosis ≥ 50% on coronary angiography
  Interventions: Device: Onyx family
- Able to take antiplatelets for at least 1 months after the procedure: Patients able to take antiplatelets after the procedure
  Interventions: Device: Onyx family
- Patients who underwent coronary artery procedures with ZES stent: Patients who underwent coronary artery procedures with Onyx™ family stent
  Interventions: Device: Onyx family

INTERVENTIONS:
Device: Onyx family — Safety and Efficacy of 1-Month DAPT in Elderly Patients at High Risk of Ischemia and Bleeding After Percutaneous Coronary Intervention with Onyx Family Stents
  Other Names: Onyx frontier; Resolute Onyx

SUMMARY:
Observation of the safety and efficacy of 1-month dual antiplatelet therapy (DAPT) after percutaneous coronary intervention using Onyx family stents in elderly patients aged 75 years or older

DETAILED DESCRIPTION:
For elderly patients aged 75 years or older undergoing percutaneous coronary intervention with Onyx family drug-eluting stents, observe the safety and efficacy of transitioning from dual antiplatelet therapy to single therapy for one year after one month of dual antiplatelet therapy

ELIGIBILITY:
Inclusion Criteria:

* Aged 75 or more.
* Eligible for interventional procedures.
* Evidence of myocardial ischemia or coronary artery stenosis ≥ 50%.
* Able to take antiplatelets for at least 1 months after the procedure.
* Patients who underwent coronary artery procedures with ZES (Medtronic, Minneapolis, MN, Onyx™ family) stent.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, zotarolimus, and contrast media (patients with documented sensitivity to contrast media which can be effectively premedicated with steroids and diphenhydramine [eg, rash] may be enrolled. Those with true anaphylaxis to prior contrast media, however, should not be enrolled).
* Patients with active pathologic bleeding.
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia).
* Noncardiac comorbid conditions are present with life expectancy <1 year or that may result in protocol noncompliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients who underwent percutaneous coronary intervention using Onyx family stents in those aged 75 years or older
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MACCE at 12 months after coronary artery intervention | 1 year after the procedure
  MACCE defined as a composite of all-cause mortality, MI, and cerebrovascular events at 12 months after the index procedure

SECONDARY OUTCOMES:
safety of procedures | 1 year after the procedure
  All-cause mortality
safety of procedures | 1 year after the procedure
  occurrence of Cardiac mortality
safety of procedures | 1 year after the procedure
  occurrence of myocardial infarction
safety of procedures | 1 year after the procedure
  occurrence of Cerebrovascular events
safety of procedures | 1 year after the procedure
  occurrence of Target vessel revascularization (TVR) event
safety of procedures | 1 year after the procedure
  occurrence of Target lesion revascularization (TLR)
safety of procedures | 1 year after the procedure
  occurrence of Stent thrombosis
safety of procedures | 1 year after the procedure
  occurrence of Bleeding Academic Research Consortium (BARC) type 2 to 5 the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Min Ku Chon, MD,PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No